CLINICAL TRIAL: NCT06087822
Title: Randomized, Double-blinded, Placebo-controlled, Multicenter Trial Investigating Performance and Safety of the Medical Device SiPore21® in Obese or Overweight Subjects With Elevated Blood Glucose Levels
Brief Title: Multicenter Trial Investigating Performance and Safety of the Medical Device SiPore21®
Acronym: SHINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sigrid Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SITH/001921
Record Dates: First submitted 2023-10-11; First posted 2023-10-18 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, multicenter clinical investigation according to Medical Device Regulation article 62
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The IMD and placebo are comparable in appearance, texture, taste, and smell, and indistinguishable in packaging and labelling, so that study participants, CRO and investigators are blinded to treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMD SiPore21® (Experimental): IMD Class IIb Total daily dose: 3 stick packs (1 x 3 main meals) uration 12 weeks
  Interventions: Device: IMD SiPore21®
- Placebo Comparator (Placebo Comparator): Placebo Total daily dose: 3 stick packs (1 x 3 main meals) duration 12 weeks
  Interventions: Device: IMD SiPore21®

INTERVENTIONS:
Device: IMD SiPore21® — The intended use/purpose to improve blood glucose control, as measured by a reduction in HbA1c

SUMMARY:
The present clinical investigation is a randomized, double-blinded, placebo-controlled, multicenter international trial, planned to be conducted in Poland, Romania and Slovakia. The investigation will be performed to establish clinical evidence regarding the performance and safety of the IMD and is aiming at evaluating the suitability of the IMD for the intended purpose and population.

DETAILED DESCRIPTION:
The proposed investigation is set out to be a randomized, double blind, placebo-controlled, multicenter study according to MDR Article 62 to investigate performance and safety of the medical device SiPore21® in subjects with obesity or overweight and elevated blood glucose levels.

The aim of this clinical investigation is to evaluate the clinical performance of the IMD for blood glucose control and its clinical safety. The endpoints selected to evaluate the effects of the IMD are based on the state-of-the-art assessments of blood glucose control (ADA, 2022).

The main hypothesis is that treatment with SiPore21® for 12 weeks will reduce the HbA1c in obese or overweight subjects with elevated blood glucose levels. It is further hypothesized that treatment with SiPore21® for 12 weeks will result in a reduction in body weight and influence metabolic control parameters and lipid levels.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-70 years old
2. HbA1c level ≥42 to 58 mmol/mol (≥6 to 7.5% - according to Diabetes Control and Complications Trial [DCCT, 1987]) at V1 For Poland only: HbA1c level ≥42 to 53 mmol/mol (≥6 to 7% - according to the Official Journal of the Diabetes Poland, 2023 Vol. 3 Issue 1) at V1
3. Body mass index (BMI) >25 kg/m2 and 40 kg/m2
4. Regular intake of 3 main meals (self-reported)
5. Readiness and ability to:

   1. use the study treatment as recommended and attend all scheduled visits
   2. comply with all further study procedures
6. Readiness to maintain the current diet and level of physical activity during the study
7. Readiness not to participate in another clinical study during this study
8. Women of childbearing potential: commitment to use medically recognized contraception methods during the treatment period
9. Written informed consent by the participant following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study

Exclusion Criteria:

1. Known allergy or hypersensitivity to the components of the IMD or placebo (self-reported)
2. Type 1 diabetes (T1D)/Latent Autoimmune Diabetes in Adult or secondary diabetes (self-reported)
3. Uncontrolled hypertension (regularly >179/109 mmHg [self-reported] and as per investigator's judgement based on screening procedures at V1)
4. History (self-reported) of myocardial infarction or stroke 6 months prior to V1
5. Clinically relevant abnormal electrocardiogram (ECG) at V1
6. History (<3 years prior to V1) or presence (self-reported) of:

   1. exocrine pancreatic insufficiency, chronic pancreatitis
   2. chronic inflammatory bowel disease, celiac disease
   3. diverticulosis (usually affecting the large intestine), adhesions, chronic constipation
7. State after pancreatic head resection with the need for additional intake of pancreatic enzymes (self-reported)
8. Major surgery of esophagus, stomach, intestine including colon which took place <3 years prior to V1, or >3 years prior to V1 in case of related current clinical symptoms (self-reported)
9. Clinically significant deviation, based on investigators judgment, in blood laboratory values at V1 of blood status (hemoglobin, erythrocytes, platelets, leucocytes, reticulocytes), kidney parameters (creatinine, cystatin C and estimated glomerular filtration rate), thyroid hormone status: thyroid-stimulating hormone (TSH)
10. Deviation in blood laboratory values at V1 of liver parameters (aspartate aminotransferase [ASAT], alanine transaminase [ALAT], alkaline phosphatase and γ-glutamyl transpeptidase [Gamma-GT]) that is clinically significant based on investigators judgment
11. Blood donation/other major blood loss or blood transfusion, that may interfere with the study as per investigator's judgment, within 56 days prior to V1 and any blood donation or transfusion during the study
12. Previous or current metformin or other medical anti-diabetic treatment or blood glucose levels reducing/influencing treatment/supplementation within 30 days prior to V1 and during the study
13. Current treatment/supplementation for weight management (e.g., fat binder/burner, carb blocker, satiety products) or known to influence weight (e.g., systemic corticosteroids)
14. Medical conditions that require medications taken during meals
15. Extreme diet form (e.g., ketogenic, very low carbohydrate) during the last 3 months prior to study
16. Self-reported regular average consumption of >1 L/day total of sugary beverages (e.g., soft drinks, fruit juices, energy drinks) and/or >200 g/day total of food based on simple sugar(s) between meals (e.g., commercial candies, dried fruit)
17. Pregnancy, lactation or active planning to achieve pregnancy
18. History of or current abuse of drugs, alcohol or medication
19. Any severe diseases/disorder (e.g., chronic kidney disease, neoplastic disease or psychiatric disorder) which may interfere with the compliance to the study procedures as per investigator's judgement
20. Participation in another study during the last 30 days prior to V1
21. Belonging to a vulnerable population, having any condition or other reason which in the opinion of the investigator would confound the conduct of the study or interpretation of the study results
22. Relative of the investigator or an employee at the clinical study site and Sponsor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or female 18-70 years old
Enrollment: 318 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
HbA1c level | Difference in changes in HbA1c levels from V2 (baseline) to V4 (week 12) between IMD treatment group and placebo group.
  To evaluate if the IMD treatment leads to a greater reduction in HbA1c level (relative to baseline) in comparison to placebo, in obese or overweight subjects with elevated blood glucose levels.

SECONDARY OUTCOMES:
Body weight | Difference in changes in body weight assessed on-site from V2 (baseline) to V4 (week 12) between IMD treatment group and placebo group.
  To evaluate if the IMD treatment leads to a greater reduction in body weight (relative to baseline) in comparison to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Klockare, Study Director — Sigrid Therapeutics
Locations (27):
- Poland (11):
  - Klimed ul. Jana Pawła II 59 lok. 6U,, Bialystok
  - RENEW Clinic ul. Gajowa 29,, Bialystok
  - Klimed Bychawa ul. Piłsudskiego 28,, Bychawa
  - Diab Serwis Popenda Spółka Jawna Józefa Ryszki 51,, Chorzów
  - Centrum Nowoczesnych Terapii Dobry Lekarz plac Szczepański 3/II,, Krakow
  - Amicare centrum medyczne Ul. Zgierska 249,, Lodz
  - Clinical Best Solutions ul. Cicha 4/1,, Lublin
  - KO-MED Centra Kliniczne Lublin II ul. K. Przerwy-Tetmajera 21, 20-362, Lublin
  - Dom Lekarski Centrum Medyczne Outlet Park ul. Andrzeja Struga 42,, Szczecin
  - MTZ Clinical Research Powered by Pratia ul. Gładka 22,, Warsaw
  - Wojskowy Szpital Kliniczny z Polikliniką SP ZOZ we Wrocławiu ul.Weigla 5,, Wroclaw
- Romania (6):
  - Neomed Strada Crișului nr. 1,, Brasov
  - Nicodiab Strada Polonă 92, Bl. 17 A+B, Bucharest
  - Spitalul Universitar de Urgenta Militar Central 'Dr Carol Davila' Calea Plevnei 134,, Bucharest
  - Fundatia Ana Aslan International Strada Vasile Pârvan, nr 12, ap 1, 010216,, Bucharest
  - RO03 MediPrax Centrum Strada Petru Maior 6-8, Cluj-Napoca
  - Clubul Sanatatii SRL Strada I. C. Brătianu 54B Cȃmpulung Muscel, Argeş, Mușcel
- Slovakia (10):
  - Metabol KLINIK, s.r.o.Cukrová 3, Bratislava
  - Metabolické centrum Dumbierska 32, Bratislava
  - DIABEDA, s.r.o.Zdravotnícke stredisko, Tbiliska 6,, Bratislava - Rača
  - Diversitas s.r.o., SNP 870/10, Hlohovec
  - INTERN, s.r.o. L. Štúra 846/39, Ilava
  - Všeobecná ambulancia pre dospelých Nábrežná 3043/3, Levice
  - SALUBER SK, s.r.o Piešťanská 1166/ 5,, Nové Mesto nad Váhom
  - MEDIPA, s.r.o., internist Sládkovicova 2A, Piešťany
  - Dr. Viliam Cibik, Pruské 293,, Pruské
  - MUDr. Dagmar Žáková Súvoz 1, Trencín

IPD SHARING:
Plan to Share IPD: No